CLINICAL TRIAL: NCT03885115
Title: Lace Up and Move: Structured After School Exercise Intervention for Hispanic and African American Youth
Brief Title: Lace Up and Move: Structured After School Intervention for Hispanic and African American Youth
Acronym: LUAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Houston (Other)
Collaborators: United Health Foundation (Unknown)
Responsible Party: Principal Investigator, Norma Olvera, Principal Investigator, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000392
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Childhood Obesity; Obesity; Physical Activity
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomly assigned to the experiential group (EG) will receive a 12-week structured exercise that will consist of two group fitness sessions (i.e. kickboxing, Zumba, fitness yoga, and other aerobic exercises) every week. Certified fitness instructors will lead each session and participants will learn strategies how to be more active during the daily routines at home. Parents or other relatives in the EG will participate in one 2-hour session every four weeks (total of 3 sessions) designed to help them support their children and entire family in being active and eat healthy at home. Parents will meet with a fitness instructor who will provide specific tips on how to increase physical activity at home as well as providing community resources to be active. A basic nutrition education and cooking demonstrations, and healthy recipes will be also provided to parents at these workshops. Data/assessments are collected, pre and post the 12 weeks intervention.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Participants randomly assigned to the control group (CG) will receive once a week recreational structured group play/game sessions led by trained BOUNCE interns/staff. The control group will receive 60 minute of structured free play sessions (i.e. recreational games) once a week for 12 weeks. Every 4 weeks, parents will be given (either sent home with their child or via email or mail) basic nutrition information, healthy recipes, and tips to promote physical activity at home as well as community resources to be active. Data/assessments are collected, pre and post the 12 weeks intervention.

INTERVENTIONS:
Behavioral: Intervention — Involves 12-weeks of education related to healthy behaviors, nutrition, and exercise from certified fitness instructors.
  Arms: Intervention

SUMMARY:
The purpose of this study is to test the efficacy of Lace Up and Move (LUAM), a structured after-school exercise intervention, designed to increase moderate-to-vigorous physical activity (MVPA) and enhance sleep quality among Hispanic and African American (AA) boys and girls.

DETAILED DESCRIPTION:
This study uses a randomized comparison-group pre-post-test design. Overall objectives of LUAM are to: (1) to increase the percentage of youth who meet 60 minutes of daily MVPA per week; (2) to improve the quality of sleep patterns (i.e., sleep efficiency and duration); and (3) to reduce percent body fat (%BF). It is hypothesized that compared to the control group (CG) participants, the experimental group (EG) participants will exhibit: (a) greater increase in percentage of children who meet 60 minutes of daily MVPA per week; (b) greater increase of sleep efficiency and duration; and (c) greater decrease in sleep latency and (d) greater decrease in %BF.

ELIGIBILITY:
Inclusion Criteria:

* child and at least their mother [or one member of the family] must be of Hispanic or African American descent
* child must have no physical disability or medical conditions that interfere with their participation in the exercise program

Exclusion Criteria:

* neither child nor parental guardians is of Hispanic or African American descent
* child is not between the ages of 9-14 years
* child is pregnant or physically unable to participate in the exercise program.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Child Physical Activity | pre & post intervention at Week 12
  measure the percentage of youth who meet 60 minutes of daily moderate-to-vigorous physical activity per week

SECONDARY OUTCOMES:
Sleep | pre & post intervention at Week 12
  assess using self-report survey
Sleep Quality | pre & post intervention at Week 12
  assess quality of sleep patterns using a small motion analyzer that measures sleep efficiency, duration and latency
Body fat percentage | pre & post intervention at Week 12
  percent body fat obtained from a foot-to-foot bio-electrical impedance assessment

CONTACTS AND LOCATIONS:
Overall Officials: Norma Olvera, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No